CLINICAL TRIAL: NCT02404324
Title: Prescription of Full Optical Correction in Refractive Errors to Treat Esotropia in Children up to 3 Years Old
Brief Title: Conservative Treatment of Esotropia in Children up to 3 Years Old
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Centre of Ophthalmology named after academician Zarifa Aliyeva (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Treatment of Esotropia
Record Dates: First submitted 2014-12-23; First posted 2015-03-31 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2015-03

CONDITIONS: Esotropia
MeSH Terms: conditions — Esotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- spectacles (Experimental): Esotropia is treated by full optical correction (spectacles prescription) in all children with refractive errors. Special attention is paid to astigmatism up to 0.5 Dptr.
  Intervention: Prescription of spectacles
  Interventions: Other: Prescription of spectacles

INTERVENTIONS:
Other: Prescription of spectacles — All children are prescribed full optical correction of refractive errors with special attention to astigmatism up to 0.5 Dptr to achieve maximal clear image on the retina of both eyes.If necessary, direct occlusion or penalization are administered to the children.

SUMMARY:
The objective of this prospective study is the treatment of esotropia by prescribing the full precise optical correction of refractive errors in children up to 3 years old.

DETAILED DESCRIPTION:
This investigation includes children with esotropia associated with hyperopia, hypermetropic astigmatism, myopia, myopic astigmatism and minor ametropias. All children are prescribed full optical correction of refractive errors with special attention to astigmatism up to 0.5 Dpt to achieve maximal clear image on the retina of both eyes.If necessary, direct occlusion or penalization were administered to the children. The investigators suggest that this approach will give good results in the treatment of esotropia.

ELIGIBILITY:
Inclusion Criteria:

* Within the age of 3 months to 3 years (inclusive infantile esotropia)
* Patients with constant or periodic esotropia and with revealed angle of deviation 5 degrees or over by Hirschberg test
* Patients with refractive errors (inclusive minor ametropias from 0.5 Dptr)

Exclusion Criteria:

* Age above 3 years
* Patients with neurological diseases and paralytic strabismus

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
The angle of deviation | 2 years
  The absolute success is defined as restored symmetrical eye position.Qualified success is considered as reduction of the angle of deviation. Patients are examined 24 months later to assess outcome of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elmar Kasimov, Professor, Study Director — National Centre of Ophthalmology named after academician Zarifa Aliyeva

IPD SHARING:
Plan to Share IPD: No